CLINICAL TRIAL: NCT00422812
Title: A Multi-center, Randomized, Double-Blind, Placebo-Controlled, Single Dose, Efficacy and Safety Outpatient Study of StaccatoTM Prochlorperazine for Inhalation in Patients With Migraine Headache
Brief Title: Staccato Prochlorperazine in Migraine (Out Patient)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-001-202
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2008-06

CONDITIONS: Migraine Headache; Aura
Keywords: Migraine, Staccato Prochlorperazine; Migraine headache with or without aura.
MeSH Terms: conditions — Migraine Disorders; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Inhaled Placebo (Placebo Comparator): Inhaled Staccato Placebo
  Interventions: Drug: Inhaled Placebo
- Inhaled PCZ 5 mg (Experimental): Inhaled Staccato Prochlorperazine 5 mg
  Interventions: Drug: Inhaled PCZ 5 mg
- Inhaled PCZ 7.5 mg (Experimental): Inhaled Staccato Prochlorperazine 7.5 mg
  Interventions: Drug: Inhaled PCZ 7.5 mg
- Inhaled PCZ 10 mg (Experimental): Inhaled Staccato Prochlorperazine 10 mg
  Interventions: Drug: Inhaled PCZ 10 mg

INTERVENTIONS:
Drug: Inhaled Placebo — Inhaled Staccato Placebo
  Arms: Inhaled Placebo
Drug: Inhaled PCZ 5 mg — Inhaled Staccato Prochlorperazine 5 mg
  Arms: Inhaled PCZ 5 mg
Drug: Inhaled PCZ 7.5 mg — Inhaled Staccato Prochlorperazine 7.5 mg
  Arms: Inhaled PCZ 7.5 mg
Drug: Inhaled PCZ 10 mg — Inhaled Staccato Prochlorperazine 10 mg
  Arms: Inhaled PCZ 10 mg

SUMMARY:
Staccato Prochlorperazine is being developed to treat patients suffering from acute migraine headaches. In October 2005, we completed a 75 patient, multi-center, double-blind placebo-controlled Phase 2A clinical trial in patients suffering from moderate to severe acute migraine headaches. This Phase 2B clinical trial of Staccato Prochlorperazine has been initiated to assess the efficacy and safety in outpatients with migraine headache with or without aura.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between the ages of 18 to 70 years, inclusive.
2. Patients who have migraine headache with or without aura (diagnosis according to International Headache Society guidelines) for at least 6 months.
3. Patients who have a history of migraine and have had at least 3 migraine attacks in the last 3 month period (but not more than 8 migraine attacks per month). Current and past migraine medication history must be recorded.
4. Patients who agree to: not use the study drug within 72 hr of a prior migraine attack, and to use the investigational medication when they have a pain rating of Moderate or Severe (on a None, Mild, Moderate or Severe Scale) prior to dosing.
5. Patients who speak, read, and understand English sufficiently well and are willing and able to provide written informed consent on an IRB approved form prior to the initiation of any study procedures.
6. Patients who are willing and able comply with the study schedule and study requirements, and agree to return to the clinic within 5 working days of use of the investigational treatment.
7. Patients who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis and in the opinion of the Principal Investigator.
8. Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study. Medically acceptable methods of contraception that may be used by the participant and/or his/her partner include abstinence, birth control pills or patches, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization and progestin implant or injection. Prohibited methods include: the rhythm method, withdrawal, condoms alone, or diaphragm alone.

Exclusion Criteria:

1. Patients who are currently taking tricyclic antidepressants, valproate, divalproex, barbitals, thiazolidinediones, phenothiazines, benzodiazepines, lithium or any hepatic toxic drugs must be excluded.
2. Patients who are currently taking medications that prolong the QT/QTc interval (see Appendix 4) must be excluded.
3. Patients with a history of contraindications to anticholinergics (bowel obstruction, urinary retention, acute glaucoma) must be excluded.
4. Patients with a history of allergy or intolerance to phenothiazines and related drugs (prochlorperazine, chlorpromazine, promethazine, mesoridazine, thioridazine, fluphenazine, perphenazine) must be excluded.
5. Patients with a history of extra-pyramidal disorders, movement disorders, neuroleptic malignant syndrome, or major affective disorder must be excluded.
6. Female patients who have a positive pregnancy test at screening or are breastfeeding must be excluded.
7. Patients who have a history within the past year of drug or alcohol dependence or abuse as defined by DSM-4 must be excluded.
8. Patients who have a history of pheochromocytoma, seizure disorder or Parkinson's disease must be excluded.
9. Patients who have a history of syncope, unstable angina, myocardial infarction (within 6 mos), congestive heart failure, or transient ischemic attack must be excluded.
10. Patients who have a history of a major neurological disorder other than migraine (subarachnoidal bleeding, stroke, brain tumor) must be excluded.
11. Patients who have any other disease(s), by history, physical examination, or laboratory abnormalities (ALT or AST > 2-fold the upper limit of normal, Bilirubin > 1.5 mg/dL, or creatinine > 1.8 mg/dL) or that in the investigator's opinion, would present undue risk to the patient or may confound the interpretation of study results must be excluded.
12. Patients who have a history of asthma or chronic obstructive lung disease should be excluded.
13. Patients who have received an investigational drug within 30 days prior to the Screening Visit must be excluded.
14. Patients who have a history of risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) must be excluded.
15. Patients who have a marked prolongation of QT/QTc interval (e.g., demonstration of a QT interval >450 ms on screening ECG) must be excluded.
16. Patients who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving prochlorperazine, or unable to use the inhalation device, must be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Spyker, PhD, MD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (25):
- United States (25):
  - Department of Neurology, Mayo Clinic, Scottsdale, Arizona
  - San Francisco Headache Clinic, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Neurological Research Institute of East Bay, Walnut Creek, California
  - Mile High Research Center, Denver, Colorado
  - Associated Neurologists of Southern Connecticut PC, Fairfield, Connecticut
  - Hartford Headache Center, Hartford, Connecticut
  - The New England Center for Headache, Stamford, Connecticut
  - MD Clinical, Hallandale, Florida
  - Palm Beach Neurological Center, West Palm Beach, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - Medvadis, Wellesley Hills, Massachusetts
  - New England Regional Headache Center, Worcester, Massachusetts
  - The Michigan Head-Pain and Neurological Institute, Ann Arbor, Michigan
  - Headache Care Center Primary Care Network, INC, Springfield, Missouri
  - Regional Clinical Research, Endwell, New York
  - Elkind Headache Center, Mount Vernon, New York
  - New York Headache Center, New York, New York
  - Island Neurological Associates, PC, Plainview, New York
  - PharmQuest, Greensboro, North Carolina
  - Health Research Associates, Cleveland, Ohio
  - ClinExcel Research, West Chester, Ohio
  - University Neurologists/OUHSC, Oklahoma City, Oklahoma
  - Houston Headache Clinic, Houston, Texas
  - Swedish Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg
Started | 98 | 104 | 93 | 105
Completed | 98 | 103 | 91 | 103
Not Completed | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg | Total
Number analyzed (Participants) | 98 | 104 | 93 | 105 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 103 | 92 | 103 | 395
  >=65 years | 1 | 1 | 1 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (12.4) | 41.7 (11.8) | 42.9 (11.3) | 40.6 (12.1) | 41.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 94 | 80 | 85 | 349
  Male | 8 | 10 | 13 | 20 | 51
Region of Enrollment [Number; unit: participants]
  United States | 98 | 104 | 93 | 105 | 400

OUTCOME MEASURES:

1. Primary Outcome: Headache Pain Relief at 2 hr
Description: Headache pain relief at 2 hr post-dose by IHS Definition (none=0 or mild=1),
Time Frame: 2 hr post-dose
Population: ITT w/ LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg
Number analyzed (Participants) | 98 | 103 | 91 | 103
Participants | 40 | 62 | 58 | 68
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled PCZ 5 mg vs Inhaled PCZ 7.5 mg vs Inhaled PCZ 10 mg; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel — Overall effect at 2 hr (by Cochran-Mantel-Haenszel) for TREATMENT

2. Secondary Outcome: Responders, Pain-Free at 2 Hours
Description: Percentage of Responders, Pain-Free, by Treatment Group over Time
Time Frame: 2 hours
Population: ITT w/ LOCF Population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg
Number analyzed (Participants) | 98 | 103 | 91 | 103
Participants | 15 | 22 | 27 | 36
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled PCZ 5 mg; Test type: Superiority; p = 0.281, Fisher Exact
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled PCZ 7.5 mg; Test type: Superiority; p = 0.0226, Fisher Exact
Statistical Analysis 3: Comparison: Inhaled Placebo vs Inhaled PCZ 10 mg; Test type: Superiority; p = 0.0019, Fisher Exact

3. Secondary Outcome: Survival of Headache Pain Relief
Description: Survival for time to the first successful headache pain relief by Pain-IHS definition over the 0 to 4 hr period by treatment assigned. Pairwise comparisons were made for each of the 3 active doses to placebo. Survival Analysis (Kaplan-Meyer) was included to evaluate treatment efficacy over the 0 to 4 hr period. All tests were 2-sided with a p-value at α=0.05.
Time Frame: 0 to 4 hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg
Number analyzed (Participants) | 103 | 91 | 103 | 98
Participants | 77 | 67 | 71 | 52
Statistical Analysis 1: Comparison: Inhaled Placebo vs Inhaled PCZ 5 mg vs Inhaled PCZ 7.5 mg vs Inhaled PCZ 10 mg; Test type: Superiority; p = 0.0007, Log Rank — Overall effect (0-4 hr) for TREATMENT by Log-rank p-value; There was no adjustment for multiple comparisons
Statistical Analysis 2: Comparison: Inhaled Placebo vs Inhaled PCZ 5 mg; Test type: Superiority; p = 0.0008, Log Rank; No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: Inhaled Placebo vs Inhaled PCZ 7.5 mg; Test type: Superiority; p = 0.0008, Log Rank — No adjustments were made for multiple comparisons
Statistical Analysis 4: Comparison: Inhaled Placebo vs Inhaled PCZ 10 mg; Test type: Superiority; p = 0.0003, Log Rank — No adjustments were made for multiple comparisons

ADVERSE EVENTS:
Time Frame: From dosing (0 hours) through 24 hours
Description: Patient self- assessment for adverse events via Patient Diary over 0-24 hours at 7 specified time points
Arm/Group | Inhaled Placebo | Inhaled PCZ 5 mg | Inhaled PCZ 7.5 mg | Inhaled PCZ 10 mg
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/104 | 0/93 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/104 | 0/93 | 0/105
Other Adverse Events (participants affected / at risk) | 12/98 | 67/104 | 67/93 | 91/105
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Placebo (N=98) | Inhaled PCZ 5 mg (N=104) | Inhaled PCZ 7.5 mg (N=93) | Inhaled PCZ 10 mg (N=105)
Fatigue (General disorders) | 3 (3) | 6 (6) | 6 (6) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3) | 9 (9)
Somnolence (Nervous system disorders) | 1 (1) | 9 (9) | 9 (9) | 6 (6)
Psychiatric Disorders (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 20 (20) | 15 (15) | 32 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 9 (9)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 6 (6) | 5 (5)
Respiratory Tract Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 4 (4) | 5 (5)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 19 (19) | 20 (20) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less